CLINICAL TRIAL: NCT00303823
Title: A Phase II Trial of Polyphenon E for Cervical Cancer Prevention
Brief Title: Green Tea Extract in Preventing Cervical Cancer in Patients With Human Papillomavirus and Low-Grade Cervical Intraepithelial Neoplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2009-00893; NCI-2009-00893 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000458081; HSC 05-40; 05-0144-01 (Other: Arizona Cancer Center - Tucson); UAZ03-1-02 (Other: DCP); P30CA023074 (NIH); N01CN35158 (NIH)
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Results first posted 2012-08-17 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2013-04

CONDITIONS: Cervical Cancer; Cervical Intraepithelial Neoplasia Grade 1; Human Papilloma Virus Infection
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections | interventions — polyphenon E

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Patients receive oral green tea extract once daily for 16 weeks in the absence of unacceptable toxicity.
  Interventions: Dietary Supplement: defined green tea catechin extract; Other: laboratory biomarker analysis
- Arm II (Placebo Comparator): Patients receive oral placebo once daily for 16 weeks in the absence of unacceptable toxicity.
  Interventions: Drug: placebo; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: placebo — Given orally
  Other Names: PLCB
  Arms: Arm II
Dietary Supplement: defined green tea catechin extract — Given orally
  Other Names: Polyphenon E
  Arms: Arm I
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial is studying green tea extract to see how well it works compared to a placebo in preventing cervical cancer in patients with human papillomavirus and low-grade cervical intraepithelial neoplasia. Chemoprevention is the use of certain substances to keep cancer from forming, growing, or coming back. The use of green tea extract may stop cervical cancer from forming in patients with human papillomavirus and low-grade cervical intraepithelial neoplasia. It is not yet known whether green tea extract is more effective than a placebo in preventing cervical cancer in patients with human papillomavirus and low-grade cervical intraepithelial neoplasia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the effect of green tea extract (Polyphenon E®) in patients with human papillomavirus (HPV) expression and low-grade cervical intraepithelial neoplasia (CIN 1) in a pre- and post-treatment setting.

SECONDARY OBJECTIVES:

I. Compare the toxicity of green tea extract vs placebo among patients with CIN 1.

TERTIARY OBJECTIVES:

I. Evaluate the utility of karyometry as an intermediate endpoint biomarker for cervical chemoprevention studies.

OUTLINE:

This is a randomized, double-blind, placebo-controlled study. Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive oral green tea extract (Polyphenon E®) once daily for 16 weeks in the absence of unacceptable toxicity.

ARM II: Patients receive oral placebo once daily for 16 weeks in the absence of unacceptable toxicity.

After completion of study treatment, patients are followed for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cervical intraepithelial neoplasia 1 (CIN 1) AND oncogenic human papillomavirus (HPV) positivity
* At increased risk for developing cervical cancer due to >= 1 of the following criteria (documented 6-12 months ago)*:

  * Positive oncogenic HPV on DNA hybrid capture
  * Low-grade squamous intraepithelial lesion cytology
  * Histopathologically documented CIN 1 on cervical biopsy [Note: *Patients must now have current CIN 1 by histology or colposcopy AND HPV positivity]
* Cervical dysplasia by colposcopy OR positive biopsy
* No invasive cervical cancer or high-grade intraepithelial neoplasia on cervical biopsy or endocervical curettage
* ECOG performance status < 2
* Total bilirubin < 2 times upper limit of normal (ULN)
* AST < 2 times ULN
* ALT normal
* Creatinine < 2.0 mg/dL
* Able and willing to return to clinic for study visits once every 4 weeks for the duration of the study
* No history of allergic reaction to tea or related dietary products
* No HIV positive patients (or AIDS/HIV-associated complex)
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection other than HPV
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situation that would limit compliance with study requirements
* No history of any cancer except nonmelanoma skin cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No regular intake of 6 or more servings of tea per week within 1 month prior to study entry
* No treatment for genital condyloma within 30 days prior to study entry
* No prior pelvic irradiation
* No concurrent tea (green, black, or oolong) or tea-derived products
* No other concurrent investigational agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2005-09; Primary Completion 2010-11 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Garcia, Principal Investigator — Arizona Cancer Center - Tucson
Locations (1):
- Arizona Cancer Center - Tucson, Tucson, Arizona, United States

REFERENCES:
- [Derived] Garcia FA, Cornelison T, Nuno T, Greenspan DL, Byron JW, Hsu CH, Alberts DS, Chow HH. Results of a phase II randomized, double-blind, placebo-controlled trial of Polyphenon E in women with persistent high-risk HPV infection and low-grade cervical intraepithelial neoplasia. Gynecol Oncol. 2014 Feb;132(2):377-82. doi: 10.1016/j.ygyno.2013.12.034. Epub 2014 Jan 2. PMID 24388920

RESULTS

PARTICIPANT FLOW:
Groups:
- Polyphenon E (Defined Green Tea Catechin Extract): Patients receive oral Polyphenon E daily for 16 weeks
- Placebo: Patients receive oral placebo once daily for 16 weeks
Period: Overall Study
Arm/Group | Polyphenon E (Defined Green Tea Catechin Extract) | Placebo
Started | 50 | 48
Completed | 35 | 38
Not Completed | 15 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Polyphenon E | Placebo | Total
Number analyzed (Participants) | 50 | 48 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 48 | 98
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.48 (8.78) | 28.27 (8.05) | 28.28 (8.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 48 | 98
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 48 | 98

OUTCOME MEASURES:

1. Primary Outcome: Complete Response - Clearance of Oncogenic Human Papillomavirus (HPV) and Complete Colposcopic, Histologic and Cytologic Clearance of Disease
Time Frame: 4 months
Measure: Number; unit: participants
Arm/Group | Polyphenon E | Placebo
Number analyzed (Participants) | 41 | 41
participants | 7 | 6

2. Primary Outcome: Partial Response - Clearance of Oncogenic HPV With Evidence of Low Grade Cervical Intraepithelial Neoplasia
Time Frame: 4 months
Measure: Number; unit: participants
Arm/Group | Polyphenon E | Placebo
Number analyzed (Participants) | 41 | 41
participants | 1 | 6

3. Primary Outcome: No Response - Persistent Oncogenic HPV Positivity, With or Without Evidence of Low Grade Cervical Intraepithelial Neoplasia
Time Frame: 4 months
Measure: Number; unit: participants
Arm/Group | Polyphenon E | Placebo
Number analyzed (Participants) | 41 | 41
participants | 27 | 26

4. Primary Outcome: Progression - Persistent Oncogenic HPV Positivity, With Evidence of Progression to Worsening Cervical Intraepithelial Neoplasia or Invasive Cancer
Time Frame: 4 months
Measure: Number; unit: participants
Arm/Group | Polyphenon E | Placebo
Number analyzed (Participants) | 41 | 41
participants | 6 | 3

ADVERSE EVENTS:
Arm/Group | Polyphenon E | Placebo
Serious Adverse Events (participants affected / at risk) | 0/50 | 1/48
Other Adverse Events (participants affected / at risk) | 42/50 | 34/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Polyphenon E (N=50) | Placebo (N=48)
Seizure (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Polyphenon E (N=50) | Placebo (N=48)
Constipation (Gastrointestinal disorders) | 2 | 4
Diarrhea (Gastrointestinal disorders) | 1 | 3
Flatulence (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 16 | 9
Vomiting (Gastrointestinal disorders) | 3 | 1
Cervicitis (Infections and infestations) | 6 | 3
Sinusitis (Infections and infestations) | 3 | 0
ALT increased (Investigations) | 5 | 1
AST increased (Investigations) | 4 | 1
Dizziness (Nervous system disorders) | 7 | 3
Fatigue (General disorders) | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Other respiratory disorders (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Irregular menses (Reproductive system and breast disorders) | 3 | 2
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 4
Other reproductive system disorders (Reproductive system and breast disorders) | 1 | 3
Abdomen pain (Gastrointestinal disorders) | 2 | 4
Stomach pain (Gastrointestinal disorders) | 6 | 4
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Other pain (General disorders) | 1 | 3
Headache (Nervous system disorders) | 13 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less